CLINICAL TRIAL: NCT04836949
Title: Verification of Shear Wave Elastography for DEtection of Prostate Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 1-2020-0072
Record Dates: First submitted 2021-04-06; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shear Wave Elastography Group (Experimental)
  Interventions: Device: Shear Wave Elastography of prostate
- Conventional ultrasonography Group (Active Comparator)
  Interventions: Device: Conventional Prostate Ultrasound

INTERVENTIONS:
Device: Shear Wave Elastography of prostate — A 12-core template biopsy is planned as during a conventional prostate biopsy. The prostate is divided in to 1) Rt apex, 2) Rt mid, 3) Rt base, 4) Rt apex lateral, 5) Rt mid lateral, 6) Rt base lateral, 7) Lt apex, 8) Lt mid, 9) Lt base, 10) Lt apex lateral, 11) Lt mid lateral, and 12) Lt base lateral areas. The elasticity of each area is evaluated and region with the maximum Young's modulus value is selected and targeted for biopsy. Additional biopsy for suspicious lesions can be performed at the discretion of the practitioner.
  Arms: Shear Wave Elastography Group
Device: Conventional Prostate Ultrasound — A conventional 12-core template biopsy is planned. The prostate is divided in to 1) Rt apex, 2) Rt mid, 3) Rt base, 4) Rt apex lateral, 5) Rt mid lateral, 6) Rt base lateral, 7) Lt apex, 8) Lt mid, 9) Lt base, 10) Lt apex lateral, 11) Lt mid lateral, and 12) Lt base lateral areas. Random biopsy of each area is performed. Additional biopsy of suspicious hypoechoic nodular lesions can be performed at the discretion of the practitioner.
  Arms: Conventional ultrasonography Group

SUMMARY:
1. Objective To provide evidence that adding shear wave elastography during sono-guided prostate biopsy can increase prostate cancer detection rate and to demonstrate that shear wave elastography of the prostate can discriminate malignant lesions to reduce the number of unnecessary prostate biopsies.
2. Overview Patients who are indicated for prostate biopsy in suspicion of prostate cancer will be assigned to a control group and an intervention group under double blinded randomization.

   * Control group : Patients will undergo prostate biopsy guided by conventional ultrasonography (B mode, gray scale).
   * Experimental group : Patients will undergo prostate biopsy guided by shear wave elastography in addition to conventional ultrasonography.

A comparative statistical analysis of the two groups will be performed.

The study is planned to be conducted for 3 years, with 2 years for patient enrollment and 1 year of follow-up. Three hospitals will participate in the study to enroll 85 patients for each group and a total of 170 patients.

3. Inclusion and Exclusion criteria

* Male patients with suspected prostate cancer must meet at least one of the following three criteria.

  1. PSA level over 4ng/dl
  2. Suspicious hard prostatic nodule on digital rectal examination.
  3. Hypoechoic lesion on ultrasound of the prostate suspicious for cancer.
* Patients who (1) are less than 20 years old, (2) have a history of surgery on the prostate such as HoLEP, (3) have moderate cognitive impairment, or (4) have medical conditions precluding transrectal procedures such as rectal cancer are excluded from the study.

  4. Research method
* Patients who wish to participate in this study and meet the inclusion/exclusion criteria are randomly assigned to the 2 groups as described above.
* The biopsy results are checked one week after the procedure.

  * Patients confirmed to have prostate cancer are provided proper treatment according to generally accepted treatment methods.
  * Patients with negative biopsy results are followed according to general follow-up protocol for suspected prostate cancer patients. After 6 months from the biopsy the patients are re-evaluated and if cancer is still suspected based on PSA level or other clinical symptoms, prostate MRI or additional biopsy is be performed.
* Patients are followed again after 12 months since the initial biopsy with identical methods from the 6 months follow-up protocol.

ELIGIBILITY:
Inclusion Criteria:

1. PSA level over 4ng/dl
2. Suspicious hard prostatic nodule on digital rectal examination.
3. Hypoechoic lesion on ultrasound of the prostate suspicious for cancer.

Exclusion Criteria:

1. Less than 20 years old
2. History of surgery on the prostate such as HoLEP
3. More than moderate cognitive impairment which limits understanding of the study
4. Medical conditions precluding transrectal procedures such as rectal cancer

Ages: 21 Years to 90 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male patients
Enrollment: 170 (Estimated)
Dates: Start 2021-05-03 (Estimated); Primary Completion 2023-12-08 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
Detection rate of prostate cancer | The presence of prostate cancer on pathologic results is checked one to two weeks after the biopsy.
  The number of subjects diagnosed with prostate cancer and the rate of detection by each group.

CONTACTS AND LOCATIONS:
Overall Officials: Woong Kyu Han, Principal Investigator — Severance Hospital
Locations (1):
- Yonsei University Health System, Severance Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No